CLINICAL TRIAL: NCT06828250
Title: Effect of Intradermal Needle Therapy for Postoperative Pain After Endoscopic Submucosal Dissection (ESD): a Prospective, Randomized Controlled Study
Brief Title: Intradermal Needle Therapy Relieves Postoperative Pain After Endoscopic Submucosal Dissection (ESD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Key Laboratory for Gastrointestinal Diseases of Gansu Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INT001
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Endoscopic Submucosal Dissection (ESD)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Both the anesthesiologist and the endoscopic surgeon involved in the procedure were blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intradermal needle therapy (Experimental): In addition to conventional treatment, patients in the treatment group received intradermal needle therapy after returning to the ward safely. Bilateral Hegu (LI4) and Zusanli (ST36) acupoints were selected for this therapy. Patients were positioned in a supine position, and after locating the acupoints, the skin of the acupoint areas was sterilized with 75% ethanol using a medical cotton swab. The intradermal needle was then removed along with the adhesive tape, inserted into the acupoints, and pressed every 4 hours for approximately 60 presses each time, excluding nighttime sleep. The pressure was applied until an acid, swelling, or numb sensation was felt at each acupoint. The intradermal needle therapy was administered only once and continuously pressed for 3 days.
  Interventions: Device: intradermal needle therapy
- conventional treatment (No Intervention): The control group received conventional postoperative treatment

INTERVENTIONS:
Device: intradermal needle therapy — In addition to conventional treatment, patients in the treatment group received intradermal needle therapy after returning to the ward safely. Bilateral Hegu (LI4) and Zusanli (ST36) acupoints were selected for this therapy. Patients were positioned in a supine position, and after locating the acupoints, the skin of the acupoint areas was sterilized with 75% ethanol using a medical cotton swab. The intradermal needle was then removed along with the adhesive tape, inserted into the acupoints, and pressed every 4 hours for approximately 60 presses each time, excluding nighttime sleep. The pressure was applied until an acid, swelling, or numb sensation was felt at each acupoint. The intradermal needle therapy was administered only once and continuously pressed for 3 days.
  Arms: intradermal needle therapy

SUMMARY:
The objective of this clinical trial is to explore the analgesic effect of intradermal needle therapy on patients after gastric endoscopic submucosal dissection； analyze factors related to postoperative pain in gastric endoscopic submucosal dissection (ESD) patients, and evaluate the safety of intradermal needle therapy.

The primary questions it aims to address are:

1. What is the incidence of moderate-to-severe pain after gastric endoscopic submucosal dissection (ESD)? What is the incidence of moderate-to-severe pain after treatment with intradermal needle therapy?
2. What adverse reactions do patients experience after treatment with intradermal needle therapy?
3. Does intradermal needle therapy alleviate postoperative pain in patients undergoing gastric endoscopic submucosal dissection (ESD)?

Patients will:

1. Postoperatively, patients were randomly assigned to a treatment group and a control group. In addition to conventional treatment, patients in the treatment group received intradermal needle therapy after returning to the ward safely. Bilateral Hegu (LI4) and Zusanli (ST36) acupoints were selected for this therapy. Patients were positioned in a supine position, and after locating the acupoints, the skin of the acupoint areas was sterilized with 75% ethanol using a medical cotton swab. The intradermal needle was then removed along with the adhesive tape, inserted into the acupoints, and pressed every 4 hours for approximately 60 presses each time, excluding nighttime sleep. The pressure was applied until an acid, swelling, or numb sensation was felt at each acupoint. The intradermal needle therapy was administered only once and continuously pressed for 3 days. The control group received conventional postoperative treatment.
2. Researchers will record the incidence of moderate-to-severe pain within 72 hours postoperatively using the VAS pain score (no pain: 0 points, mild: 1-3 points, moderate: 4-6 points, severe: 7-10 points). VAS pain scores and Simplified McGill Pain Questionnaire (SF-MPQ) scores will be assessed upon safe return to the ward, at 6h, 12h, 24h, 48h, and 72h postoperatively. The use of analgesic medications will also be noted. Preoperative and postoperative SAS and SDS scores will be documented, along with postoperative recovery details such as length of hospital stay and time of first flatus after surgery, and surgical complications (such as fever, bleeding, and perforation). Additionally, the safety evaluation of intradermal needle therapy will include monitoring for adverse events such as dizziness, skin irritation, skin breakage, infection, hematoma, local pain or discomfort at the puncture site, or needle breakage.
3. The baseline characteristics of patients will be recorded, and factors associated with postoperative pain after gastric endoscopic submucosal dissection (ESD) (including demographic data, clinicopathological features, surgical conditions, etc.) will be analyzed.

DETAILED DESCRIPTION:
Objective: To investigate the analgesic effect and safety of intradermal needle therapy for patients after gastric endoscopic submucosal dissection (ESD).

Methods: Patients undergoing gastric endoscopic submucosal dissection (ESD) treatment at a digestive endoscopy center in Lanzhou, Gansu Province, starting in January 2025, were selected as the subjects of this study.

1. Research Design: Inclusion and exclusion criteria for patients undergoing gastric endoscopic submucosal dissection (ESD) were established for screening purposes. Selected patients signed informed consent forms. Following endoscopic submucosal dissection (ESD) , patients were randomly divided into a treatment group and a control group at a 1:1 ratio based on a random number table. The treatment group received intradermal needle therapy in addition to conventional treatment, administered uniformly by trained nursing staff. The control group received conventional treatment only. Both the anesthesiologist and the endoscopic surgeon involved in the procedure were blinded to the group allocation. However, due to the particularity of the intradermal needle therapy, it was not possible to blind the patients.
2. Data collection: Patient demographic data (age, gender, height, weight, comorbidities, smoking, and drinking status), clinicopathological characteristics (location, depth, and pathological classification), and surgery-related information (duration of surgery, surgery-related complications) were collected. Additionally, the occurrence of nausea, vomiting, and abdominal distension during the trial, the location of pain, and the levels of white blood cells and C-reactive protein on the first postoperative day were recorded.
3. Outcomes: The primary outcome of the clinical trial was the incidence of moderate-to-severe pain within 72 hours postoperatively. Secondary outcomes included VAS pain scores at various time points (immediately after returning safely to the ward, 6h, 12h, 24h, 48h, and 72h postoperatively), Simplified McGill Pain Score (SF-MPQ), use of analgesic medications, preoperative and postoperative SAS and SDS scores, postoperative recovery status (including hospital stay duration and time of first postoperative flatulence), surgical complications (such as fever, bleeding, and perforation), and safety evaluation of intradermal needle therapy (including adverse reactions such as dizziness, skin allergy, skin damage, infection, hematoma, local pain, or other discomforts at the puncture site, or needle breakage).
4. Sample Size Calculation: The sample size calculation was based on the findings from a preliminary experiment, where the incidence of moderate-to-severe postoperative pain was 10% in the treatment group and 40% in the control group. This difference was used to calculate the required sample size to detect clinically significant differences between the groups using PASS.2021 software. With a type 1 error probability of 0.05 (α = 0.05), a type 2 error probability of 0.2 (β = 0.2), and a power of 0.80 for a two-sided comparison and based on the aforementioned between-group difference in the incidence of moderate-to-severe postoperative pain, we determined that 64 patients were required in each group. Accounting for a 20% lost-to-follow-up rate and a 1:1 enrollment ratio, a total sample size of 78 patients (39 in each group) was included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the surgical indications for gastric endoscopic submucosal dissection;
2. All patients signed a written "Surgical Consent Form" before surgery;
3. Complete clinical data;
4. Informed consent and participation in this study.

Exclusion Criteria:

1. Patients who have been taking oral analgesic drugs chronically before surgery;
2. Patients with severe cardiac, liver, or kidney dysfunction, or coagulation abnormalities;
3. Exclusion of patients with cardiogenic chest pain;
4. Individuals with psychiatric disorders, impaired communication abilities, or difficulties in self-assessment of pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of moderate-to-severe pain within 72 hours postoperatively | 72 hours postoperatively
  the VAS pain score (no pain: 0 points, mild: 1-3 points, moderate: 4-6 points, severe: 7-10 points).

IPD SHARING:
Plan to Share IPD: No